CLINICAL TRIAL: NCT06178497
Title: 5 Years' Follow-up Assessment of Surgical Repair for ACL Proximal Rupture
Acronym: RUPTUPROX
Status: Recruiting | Type: Observational
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Other Study IDs: RGDS-2023-06-043
Record Dates: First submitted 2023-12-11; First posted 2023-12-21 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: ACL - Anterior Cruciate Ligament Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Isolated ruptures of ACL (anterior cruciate ligament) are ligament injuries that can be proximal, central or distal. Treatment of patients with proximal lesions should be graded. Functional treatment can be reserved for low-demanding patients in whom the practice level is limited and progression risk to a functionally unstable knee less marked. In athletes, the risk of a new sprain must be explained and the patient will choose functional treatment or surgical treatment.

Surgical treatment generally involves ligamentoplasty at the expense of a knee tendon to replace the ruptured ACL. In the context of proximal ACL rupture, the patient can be offered surgical repair of the ACL. There are numerous studies on ACL ligamentoplasties results but literature is poor on modern ACL repair outcomes.

In this context, this study aims to describe the relapse rate at 5 years of patients operated for a proximal ACL tear.

DETAILED DESCRIPTION:
Isolated ruptures of ACL (anterior cruciate ligament) are ligament injuries which lead to the most surgical interventions on the capsuloligamentous system of the knee. These ruptures can be proximal, central or distal.

Treatment of patients with proximal lesions should be graded and should take into account the patient's symptoms (feeling of instability), physical examination data, amount of residual ligament, sport practice, practice level, interval time since the initial trauma, work requirements… Functional treatment can be reserved for low-demanding patients in whom the practice level is limited and tprogression risk to a functionally unstable knee less marked. In athletes, the risk of a new sprain must be explained and the patient will choose functional treatment or surgical treatment.

Functional treatment is variable, combining the use of splints, rehabilitation, muscle strengthening. The healing time is three months. Wearing a splint has not proven its effectiveness in preventing progression to complete rupture when resuming sport activities. If instability is revealed, it is then necessary to move towards ACL reconstruction treatment.

Surgical treatment generally involves ligamentoplasty at the expense of a knee tendon to replace the ruptured ACL. In the context of proximal ACL rupture, the patient can also be offered surgical repair of the ACL. There are numerous studies on ACL ligamentoplasties results but literature is poor on modern ACL repairs outcomes. Surgical repair of proximal rupture of ACL has experienced renewed interest in recent years thanks to the appearance of new fixing systems. Used in the 1980s, this technique was gradually abandoned in the mid-1980s following disappointing results for the benefit of autograft reconstruction techniques.

Few studies exist in the literature on long-term ACL repair surgery follow-up. In this context, this study aims to describe the relapse rate at 5 years of patients operated for a proximal ACL tear.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, aged ≥ 18 years
* Patient with no history of knee surgery except meniscal surgery
* Patient with an isolated proximal Sherman 1 or 2 ACL tear
* Patient with a proximal Sherman 1 or 2 ACL tear associated to a meniscal lesion
* Patient with a proximal ACL tear associated with an injury to the MCL or LCL grade 1 or 2 but not grade 3
* Patient whose period is less than 3 months between the date of the accident and the surgery
* Patient who received surgical repair between January 2019 and July 2021

Exclusion Criteria:

* Patient with contralateral ACL tear
* Patient with ACL tear Sherman 3 or 4
* Patient with a surgical history on the knee concerned, other than meniscal surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a 5 years MRI follow up after proximal ACL tear repair
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
ACL rupture relapse rate | 1 day
  ACL rupture relapse will be assessed on MRI 5 years after ACL surgery

CONTACTS AND LOCATIONS:
Overall Officials: Romain LETARTRE, MD, Principal Investigator — Hôpital Privé La Louvière
Locations (1):
- Hôpital Privé La Louvière, Lille, Choisir Une Région, France

IPD SHARING:
Plan to Share IPD: No